CLINICAL TRIAL: NCT06953141
Title: Ultrasound Use to Estimate the Amount of Intra-abdominal Blood Following Gynecological Surgeries and the Association With Postoperative Outcomes. A Prospective Cohort Study
Brief Title: Ultrasound for Assessment of Intra-Abdominal Blood Loss After Gynecological Surgery
Status: Recruiting | Type: Observational
Sponsor: Holy Family Hospital, Nazareth, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, Head of Obstetrics and Gynecology Department, Holy Family Hospital, Nazareth, Israel
Other Study IDs: 308-2025-HFH
Record Dates: First submitted 2025-04-19; First posted 2025-05-01 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Post-Operative Hematoma at Operative Site (Diagnosis); Post-Operative Hemorrhage
MeSH Terms: conditions — Disease; Postoperative Hemorrhage | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Abdominal and transvaginal ultrasound
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Transabdominal and transvaginal imaging will be performed to eligible women following gynecological surgery within 24 - 48 hours.

SUMMARY:
This is a prospective cohort study designed to assess intra-abdominal blood volume and hemodynamic status by measuring the diameter of the inferior vena cava (IVC) using 3D and Doppler ultrasound within 24 hours after gynecological surgery. The study will examine the association between these ultrasound findings and postoperative outcomes, including hemoglobin drop, need for blood transfusion, pain, infection, and length of hospitalization. Approximately 250 women undergoing laparotomy, laparoscopy, or vaginal surgery at Holy Family Hospital will be enrolled. The study also aimed to define postoperative normograms for fluid volume and IVC parameters and to evaluate whether ultrasound-guided decision-making could improve postoperative care and reduce unnecessary interventions.

DETAILED DESCRIPTION:
Postoperative intra-abdominal bleeding is a significant contributor to morbidity and, in some cases, mortality following gynecological surgery. Timely recognition of intra-abdominal blood loss is essential for appropriate clinical intervention. In cases where bleeding is into the abdominal cavity, diagnosis is more difficult and may be delayed.

Ultrasound is a non-invasive, rapid, and widely available tool for assessing free intra-abdominal and pelvic fluid. Modern machines allow for 3D volumetric assessment of fluid collections, as well as Doppler-based measurements of the inferior vena cava (IVC) diameter and its collapsibility index-both of which are known to correlate with intravascular volume status and blood loss. Currently, there are limited data establishing normal ranges of intra-abdominal fluid or IVC diameter postoperatively, and little is known about the magnitude of these measurements and clinical outcomes after gynecologic procedures.

This prospective cohort study aims to quantify intra-abdominal fluid and determine IVC diameter and its collapsibility index using advanced ultrasound imaging within 24 hours after surgery. Patients undergoing open, laparoscopic, or vaginal gynecological procedures will be included. The study will explore correlations between ultrasound findings and clinical outcomes such as hemoglobin drop, need for blood transfusion, infection, pain, and length of hospital stay. Additionally, we aim to develop reference normograms for postoperative normal ranges of intraabdominal fluid volume and IVC diameter.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Undergoing gynecological surgery including laparotomy, laparoscopy, and vaginal pelvic surgery
* Able to provide informed consent

Exclusion Criteria:

* Undergoing minor procedures (e.g., dilation and curettage, hysteroscopy, or cervical conization)
* Known preoperative coagulation disorders
* Postoperative admission to the intensive care unit (ICU)
* Clinical indication requiring ultrasound as part of standard postoperative care

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years and older undergoing gynecological surgery (open, laparoscopic, or vaginal) at Holy Family Hospital in Nazareth, Israel.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of intra-abdominal free fluid | Within 24-48 hours after surgery
  Detection of any intra-abdominal or pelvic free fluid via ultrasound examination within 24 - 48 hours after gynecological surgery.

SECONDARY OUTCOMES:
Volume of intra-abdominal fluid | Within 24-48 hours after surgery
  Measured in mL using 3D ultrasound
Presence and size of pelvic hematoma | Within 24-48 hours after surgery
  Using ultrasound to identify hematomas and measure their volume
Inferior vena cava (IVC) diameter and collapsibility index | Within 24-48 hours after surgery
  Using ultrasound Doppler to measure Inferior vena cava (IVC) diameter and collapsibility index
Hemoglobin drop | Within 24-48 hours after surgery
  Delta hemoglobin level before surgery and at 48-72 hours postoperatively.
Need for blood transfusion | Within 72 hours after surgery
  Number of packed red blood cells administered during hospitalization.
Length of hospital stay | Day 1 to day 7 after operation
  Total duration of hospitalization in days.
Surgical site infection | Within 96 hours after surgery
  Recording any infection in the part of the body where a surgery took place
Postoperative fever | Within 96 hours after surgery
  Body temperature ≥38.0°C within 72 hours after surgery.
Patient discomfort from the ultrasound examination | Immediately after ultrasound examination
  Measured on a scale of 1 to 5 (1 = no discomfort, 5 = very uncomfortable).

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Study Chair — Holy Family Hospital, Nazareth, Israel
Locations (1):
- Holy Family hospital, Nazareth, Nazareth, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Massalha M, Faranish R, Romano S, Salim R. Decreased inferior vena cava diameter as an early marker in postpartum hemorrhage. Ultrasound Obstet Gynecol. 2022 Feb;59(2):234-240. doi: 10.1002/uog.23695. Epub 2022 Jan 18. PMID 34076923
- [Background] Faustin D, Minkoff H, Schaffer R, Crombleholme W, Schwarz R. Relationship of ultrasound findings after cesarean section to operative morbidity. Obstet Gynecol. 1985 Aug;66(2):195-8. PMID 3895070
- [Background] Naeiji Z, Sotudeh S, Keshavarz E, Naghshvarian N, Rahmati N. Risk factors and clinical significance of abdomino-pelvic free fluid after cesarean section: a prospective study. J Matern Fetal Neonatal Med. 2021 Jan;34(2):287-292. doi: 10.1080/14767058.2019.1605351. Epub 2019 May 15. PMID 30957592
- [Background] Antonelli E, Morales MA, Dumps P, Boulvain M, Weil A. Sonographic detection of fluid collections and postoperative morbidity following Cesarean section and hysterectomy. Ultrasound Obstet Gynecol. 2004 Apr;23(4):388-92. doi: 10.1002/uog.1023. PMID 15065191
- [Background] Hoppenot C, Tankou J, Stair S, Gossett DR. Sonographic evaluation for intra-abdominal hemorrhage after cesarean delivery. J Clin Ultrasound. 2016 May;44(4):240-4. doi: 10.1002/jcu.22289. Epub 2015 Aug 24. PMID 26302357
- [Background] Dane C, Dane B, Cetin A, Yayla M. Sonographically diagnosed vault hematomas following vaginal hysterectomy and its correlation with postoperative morbidity. Infect Dis Obstet Gynecol. 2009;2009:91708. doi: 10.1155/2007/91708. Epub 2007 Feb 28. PMID 17485823